CLINICAL TRIAL: NCT04615273
Title: foresiGHt: A Multicenter, Randomized, Parallel-arm, Placebo-controlled (Double- Blind) and Active-controlled (Open-label) Trial to Compare the Efficacy and Safety of Once-weekly Lonapegsomatropin With Placebo and a Daily Somatropin Product in Adults With Growth Hormone Deficiency
Brief Title: A Trial to Compare the Efficacy and Safety of Once-weekly Lonapegsomatropin With Placebo and a Daily Somatropin Product in Adults With Growth Hormone Deficiency
Acronym: foresiGHt
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Ascendis Pharma Endocrinology Division A/S (Industry)
Responsible Party: Sponsor
Organization: Ascendis Pharma A/S (Industry)
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: TCH-306; 2020-000929-42 (EudraCT Number)
Record Dates: First submitted 2020-10-29; First posted 2020-11-04 (Actual); Results first posted 2025-01-15 (Actual); Last update posted 2025-01-15 (Actual); Status verified 2024-12

CONDITIONS: Growth Hormone Deficiency; Endocrine System Diseases; Hormone Deficiency
Keywords: Human Growth Hormone; hGH; rhGH; GHD; Adult Growth Hormone Deficiency; Long-Acting Growth Hormone; Lonapegsomatropin; Prodrug; Growth Failure; Growth Hormone Replacement Therapy; Sustained Release Growth Hormone; Growth Hormone Deficiency; TransCon hGH
MeSH Terms: conditions — Dwarfism, Pituitary; Endocrine System Diseases; Failure to Thrive | interventions — lonapegsomatropin; Human Growth Hormone

STUDY DESIGN:
Intervention Model Description: Double-blind, placebo-controlled, parallel group with participants randomized into 3 treatment groups (1:1:1); lonapegsomatropin once-weekly, placebo for lonapegsomatropin once-weekly, somatropin daily.
Who Masked: Participant, Investigator
Masking Description: Once-weekly lonapegsomatropin and once-weekly placebo treatment arms were double-blinded, daily somatropin product was open-label.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (3):
- Lonapegsomatropin (Experimental): Lonapegsomatropin administered once-weekly by subcutaneous injection.
  Interventions: Drug: Lonapegsomatropin
- Placebo (Placebo Comparator): Placebo for Lonapegsomatropin administered once-weekly by subcutaneous injection.
  Interventions: Other: Placebo
- Somatropin (Active Comparator): Somatropin administered once-daily by subcutaneous injection.
  Interventions: Drug: Somatropin

INTERVENTIONS:
Drug: Lonapegsomatropin — Due to the different human growth hormone (hGH) dose requirements, depending on participant's age and concomitant use of oral estrogen, this trial has 3 dosing groups per arm, followed by gradual increasing dose titration to a target maintenance dose.
  Arms: Lonapegsomatropin
Other: Placebo — The placebo for lonapegsomatropin drug product contained the same excipients as lonapegsomatropin drug product but does not contain lonapegsomatropin itself. The placebo solution was administered by subcutaneous (SC) injection via syringe and needle. Due to the different hGH dose requirements, depending on participant's age and concomitant use of oral estrogen, this trial has 3 dosing groups and the placebo received the same dose volume as if they were randomized to once-weekly lonapegsomatropin.
  Arms: Placebo
Drug: Somatropin — Somatropin solution is provided in a pre-filled pen intended for daily subcutaneous injection. Due to the different hGH dose requirements, depending on participant's age and concomitant use of oral estrogen, this trial has 3 dosing groups per arm, followed by gradual increasing dose titration to a target maintenance dose.
  Arms: Somatropin

SUMMARY:
A 38-week dosing trial of lonapegsomatropin, a long-acting growth hormone product, administered once-a-week versus placebo-control. A daily somatropin product arm is also included to assist clinical judgement on the trial results. A total of 264 adults (males and females) with growth hormone deficiency were included. Randomization occurred in a 1:1:1 ratio (lonapegsomatropin: placebo: daily somatropin product). This is a global trial conducted in, but not limited to, the United States, Europe, and Asia.

ELIGIBILITY:
Inclusion Criteria

1. Age between 23 and 80 years, inclusive, at screening.
2. Adult Growth Hormone Deficiency (AGHD) Diagnosis Criteria

   * For adult-onset AGHD: documented history of structural hypothalamic-pituitary disease, hypothalamic-pituitary surgery, cranial irradiation, 1-4 non-GH pituitary hormone deficiencies, a proven genetic cause of GHD, or traumatic brain injury (TBI).
   * Participants with childhood-onset GHD must have had GH axis re-assessed at final height.
   * In participants with TBI as a cause of GHD, GHD must be confirmed by GH -stimulation testing performed at least 12 months after the injury.

   A. For all countries except Japan: participants must have satisfied at least one of the following criteria:
   1. Insulin tolerance test: peak growth hormone (GH) <=5 ng/mL
   2. Glucagon stimulation test according to body mass index (BMI)

      * i. BMI <=30 kg/m^2: peak GH <=3 ng/mL
      * ii. BMI >30 kg/m^2: peak GH <=1 ng/mL
   3. Three or four pituitary axis deficiencies (i.e., adrenal, thyroid, gonadal, and/or vasopressin; not including GH) with insulin-like growth factor-1 standard deviation score (IGF-1 SDS) <= -2.0 at screening
   4. Macimorelin test: peak GH <=2.8 ng/mL
   5. Growth hormone releasing hormone (GHRH) + arginine test according to BMI:

      * i. BMI <25 kg/m^2, peak GH <11 ng/mL
      * ii. BMI >=25-<=30 kg/m^2, peak GH <8 ng/mL
      * iii. BMI >30 kg/m^2, peak GH <4 ng/mL

   B. For Japan only: Participants with AGHD and deficiency of at least one non-GH pituitary hormones need to satisfy one of the following GH stimulation tests. Participants with GHD without additional non-GH pituitary hormone deficiencies with or without and evidence of intracranial structure disorder need to satisfy at least 2 of the following stimulation tests:
   1. Insulin tolerance test: peak GH <=1.8 ng/mL
   2. Glucagon test: peak GH <=1.8 ng/mL
   3. Growth Hormone Releasing Peptide-2 (GHRP-2) tolerance test: peak GH <=9 ng/mL
3. IGF-1 SDS <= -1.0 at screening as measured by central laboratory.
4. hGH treatment naïve or no exposure to hGH therapy or GH secretagogue for at least 12 months prior to screening.
5. For participants on hormone replacement therapies for any hormone deficiencies other than GH (e.g., adrenal, thyroid, estrogen, testosterone) must be on adequate and stable doses for >=6 weeks prior to and throughout screening.
6. For participants not on glucocorticoid replacement therapy, documentation of adequate adrenal function at screening defined as: morning (6:00-10:00 AM) serum cortisol >15.0 mcg/dL (measured at central laboratory) and/or adrenocorticotropic hormone (ACTH) stimulation test or insulin tolerance test with serum cortisol >18.0 mcg/dL at or within 90 days prior to screening.
7. For males not on testosterone replacement therapy: morning (6:00 - 10:00AM) total testosterone within normal limits for age.
8. On a stable diet and exercise regime at screening with no intention to modify diet or exercise pattern during the trial, i.e., no weight reduction program intended during the trial or within the last 90 days prior to or through screening.
9. No plans to undergo bariatric surgery during the trial.
10. Fundoscopy at screening without signs/symptoms of intracranial hypertension or diabetic retinopathy above stage 2 / moderate or above or any other retinal disease contraindicated to growth hormone therapy. For participants with a diagnosis of diabetes mellitus at screening, this must be documented with a fundus photograph.
11. Able and willing to provide a written informed consent and authorization for protected health information (PHI) disclosure in accordance with Good Clinical Practice (GCP).
12. Serum free thyroxine (fT4) in the normal range at screening as measured by central laboratory.

Exclusion Criteria

1. Known Prader-Willi Syndrome and/or other genetic diseases that may have an impact on an endpoint.
2. Diabetes mellitus at screening if any of the following criteria are met:

   1. Poorly controlled diabetes, defined as HbA1c >7.5% at screening.
   2. Diabetes mellitus (defined as HbA1c >=6.5% and/or fasting plasma glucose >=126 mg/dL and/or plasma glucose >=200 mg/dL two hours after oral glucose tolerance test) diagnosed <26 weeks prior to screening
   3. Change in diabetes regimen (includes dose adjustment) within <90 days prior and throughout screening
   4. Use of any diabetes drugs other than metformin and/or dipeptidyl peptidase-4 (DPP-4) inhibitors for a cumulative duration of greater than 4 weeks within 12 months prior to screening
   5. Diabetes-related complications at screening (i.e., nephropathy as judged by the investigator, neuropathy requiring pharmacological treatment, retinopathy stage 2/moderate and above within 90 days prior to screening or during screening)
3. Active malignant disease or history of malignancy. Exceptions to this exclusion criterion:

   1. Resection of in situ carcinoma of the cervix uteri
   2. Complete eradication of squamous cell or basal cell carcinoma of the skin
   3. Participants with GHD attributed to treatment of intracranial malignant tumors or leukemia, provided that a recurrence-free survival period of at least 5 years prior to screening is documented in the participant's file (based on a Magnetic Resonance Imaging (MRI) result for intracranial malignant tumors)
4. Evidence of growth of pituitary adenoma or other benign intracranial tumor within the last 12 months before screening.
5. Participants with acromegaly without remission / with documented remission less than 24 months prior to screening.
6. Participants with Cushing's disease without remission / with documented remission less than 24 months prior to screening.
7. Participants with prior cranial irradiation or hypothalamic-pituitary surgery: the procedure was to take place less than 12 months prior to screening.
8. Estimated glomerular filtration rate (eGFR) <60 mL/min/1.73m^2 determined based on Modification of Diet in Renal Disease (MDRD) equation.
9. Hepatic transaminases (i.e., aspartate aminotransferase [AST] or alanine aminotransferase [ALT]) >3 times the upper limit of normal.
10. Heart failure New York Heart Association (NYHA) class 3 or greater (NYHA 1994).
11. Q-T interval, corrected by Fridericia's method (QTcF) >= 451 milliseconds on 12-lead electrocardiogram (ECG) at screening.
12. Poorly controlled hypertension, defined as supine systolic blood pressure >159 mmHg and/or supine diastolic blood pressure >95 mmHg at screening.
13. Cerebrovascular accident within 5 years prior to screening.
14. Anabolic steroids (other than gonadal steroid replacement therapy) or oral/intravenous/intramuscular corticosteroids within 90 days prior to or throughout screening.
15. Currently using or have used within 26 weeks prior to screening any weight-loss or appetite-suppressive medications including orlistat, zonisamide, lorcaserin, bupropion, topiramate, sibutramine, stimulants, glucagon-like peptide 1 (GLP-1) receptor agonists, sodium-dependent glucose cotransporters (SGLT-2) inhibitors or medications that affects IGF-1 or GH measurements including cabergoline at doses above 0.5 mg weekly or bromocriptine at doses above 20 mg weekly.
16. Known history of hypersensitivity and/or idiosyncrasy to any of the test compounds (somatropin) or excipients employed in this trial.
17. Known history of neutralizing anti-hGH antibodies.
18. Inability to undergo scanning by dual-energy x-ray absorptiometry (DXA) or a non-interpretable DXA scan at screening.
19. Female who is pregnant, breast-feeding or intends to become pregnant or is of childbearing potential (i.e., fertile, following menarche and until becoming post-menopausal unless permanently sterile) and not using adequate contraceptive methods.
20. Male participants must use a condom, or his female partner of childbearing potential must use an effective form of contraception as described above, from the beginning of screening to the last trial visit.
21. Known substance abuse or known (or previous) eating disorders, including anorexia nervosa, bulimia and severe gastrointestinal disease affecting normal eating (as judged by the investigator).
22. Any disease or condition that, in the judgement of the investigator, may make the subject unlikely to comply with the requirements of the trial or any condition that presents undue risk from the investigational product or procedures.
23. Participation in another interventional clinical trial involving an investigational compound within 26 weeks prior to screening or in parallel to this trial.
24. Currently using or have used within the last 3 days prior to screening: biotin >0.03 mg/day from supplements
25. Known history of positive results of tests for human immunodeficiency virus (HIV) antibodies or hepatitis B and/or C (exceptions if vaccinated towards Hepatitis B virus and Hepatitis C virus).
26. Any of the following: acute critical illness, and complications following open heart surgery, abdominal surgery, multiple accidental traumas, acute respiratory failure, or similar conditions within 180 days prior to screening.

Ages: 23 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 264 (Actual)
Dates: Start 2020-12-03 (Actual); Primary Completion 2023-11-02 (Actual); Study Completion 2023-12-01 (Actual)

CONTACTS AND LOCATIONS:
Locations (102):
- United States (21):
  - Ascendis Pharma Investigational Site, Birmingham, Alabama
  - Ascendis Pharma Investigational Site, Phoenix, Arizona
  - Ascendis Pharma Investigational Site, Fresno, California
  - Ascendis Pharma Investigational Site, Los Angeles, California
  - Ascendis Pharma Investigational Site, Palo Alto, California
  - Ascendis Pharma Investigational Site, Torrance, California
  - Ascendis Pharma Investigational Site, Chicago, Illinois
  - Ascendis Pharma Investigational Site, Indianapolis, Indiana
  - Ascendis Pharma Investigational Site, Boston, Massachusetts
  - Ascendis Pharma Investigational Site, Dearborn, Michigan
  - Ascendis Pharma Investigational Site, Rochester, Minnesota
  - Ascendis Pharma Investigational Site, St Louis, Missouri
  - Ascendis Pharma Investigational Site, Las Vegas, Nevada
  - Ascendis Pharma Investigational Site, Reno, Nevada
  - Ascendis Pharma Investigational Site, New York, New York
  - Ascendis Pharma Investigational Site, Morehead City, North Carolina
  - Ascendis Pharma Investigational Site, Portland, Oregon
  - Ascendis Pharma Investigational Site, Pittsburgh, Pennsylvania
  - Ascendis Pharma Investigational Site, Dallas, Texas
  - Ascendis Pharma Investigational Site, San Antonio, Texas
  - Ascendis Pharma Investigational Site, Seattle, Washington
- Ascendis Pharma Investigational Site, Yerevan, Armenia
- Australia (6):
  - Ascendis Pharma Investigational Site, Saint Leonards, New South Wales
  - Ascendis Pharma Investigational Site, Sydney, New South Wales
  - Ascendis Pharma Investigational Site, Box Hill, Victoria
  - Ascendis Pharma Investigational Site, Fitzroy, Victoria
  - Ascendis Pharma Investigational Site, Parkville, Victoria
  - Ascendis Pharma Investigational Site, Perth, Western Australia
- Canada (2):
  - Ascendis Pharma Investigational Site, Vancouver, British Columbia
  - Ascendis Pharma Investigational Site, Halifax, Nova Scotia
- Ascendis Pharma Investigational Site, Copenhagen, Denmark
- France (4):
  - Ascendis Pharma Investigational Site, Lyon
  - Ascendis Pharma Investigational Site, Marseille
  - Ascendis Pharma Investigational Site, Nantes
  - Ascendis Pharma Investigational Site, Paris
- Ascendis Pharma Investigational Site, Tbilisi, Georgia
- Ascendis Pharma Investigational Site, München, Bavaria, Germany
- Greece (3):
  - Ascendis Pharma Investigational Site, Athens, Attica
  - Ascendis Pharma Investigational Site, Thessaloniki, Central Macedonia
  - Ascendis Pharma Investigational Site, Thessaloniki
- Israel (4):
  - Ascendis Pharma Investigational Site, Beersheba
  - Ascendis Pharma Investigational Site, Haifa
  - Ascendis Pharma Investigational Site, Petah Tikva
  - Ascendis Pharma Investigational Site, Tel Aviv
- Italy (3):
  - Ascendis Pharma Investigational Site, Genova
  - Ascendis Pharma Investigational Site, Rome
  - Ascendis Pharma Investigational Site, Rozzano
- Japan (16):
  - Ascendis Pharma Investigational Site, Kobe, Hyōgo
  - Ascendis Pharma Investigational Site, Kawasaki, Kanagawa
  - Ascendis Pharma Investigational Site, Yokohama, Kanagawa
  - Ascendis Pharma Investigational Site, Matsumoto, Nagano
  - Ascendis Pharma Investigational Site, Kashihara, Nara
  - Ascendis Pharma Investigational Site, Ishikawa, Okinawa
  - Ascendis Pharma Investigational Site, Suita, Osaka
  - Ascendis Pharma Investigational Site, Chiba
  - Ascendis Pharma Investigational Site, Fukuoka
  - Ascendis Pharma Investigational Site, Kagoshima
  - Ascendis Pharma Investigational Site, Kawasaki
  - Ascendis Pharma Investigational Site, Nagakute
  - Ascendis Pharma Investigational Site, Okayama
  - Ascendis Pharma Investigational Site, Osaka
  - Ascendis Pharma Investigational Site, Tokyo
  - Ascendis Pharma Investigational Site, Yamagata
- Malaysia (4):
  - Ascendis Pharma Investigational Site, George Town
  - Ascendis Pharma Investigational Site, Kota Bharu
  - Ascendis Pharma Investigational Site, Malacca
  - Ascendis Pharma Investigational Site, Putrajaya
- Ascendis Pharma Investigational Site, Leiden, Netherlands
- New Zealand (2):
  - Ascendis Pharma Investigational Site, Palmerston North, Manawatu-Wanganui
  - Ascendis Pharma Investigational Site, Wellington
- Poland (5):
  - Ascendis Pharma Investigational Site, Krakow
  - Ascendis Pharma Investigational Site, Lodz
  - Ascendis Pharma Investigational Site, Poznan
  - Ascendis Pharma Investigational Site, Warsaw
  - Ascendis Pharma Investigational Site, Wroclaw
- Romania (3):
  - Ascendis Pharma Investigational Site, Bucharest
  - Ascendis Pharma Investigational Site, Iași
  - Ascendis Pharma Investigational Site, Timișoara
- Serbia (2):
  - Ascendis Pharma Investigational Site, Belgrade
  - Ascendis Pharma Investigational Site, Kragujevac
- Slovakia (2):
  - Ascendis Pharma Investigational Site, Bratislava
  - Ascendis Pharma Investigational Site, Ľubochňa
- South Korea (2):
  - Ascendis Pharma Investigational Site, Seoul
  - Ascendis Pharma Investigational Site, Suwon
- Spain (5):
  - Ascendis Pharma Investigational Site, Alicante
  - Ascendis Pharma Investigational Site, Barcelona
  - Ascendis Pharma Investigational Site, Madrid
  - Ascendis Pharma Investigational Site, Santiago de Compostela
  - Ascendis Pharma Investigational Site, Seville
- Turkey (Türkiye) (6):
  - Ascendis Pharma Investigational Site, Ankara
  - Ascendis Pharma Investigational Site, Antalya
  - Ascendis Pharma Investigational Site, Aydin
  - Ascendis Pharma Investigational Site, Izmir
  - Ascendis Pharma Investigational Site, İzmit
  - Ascendis Pharma Investigational Site, Kayseri
- Ukraine (4):
  - Ascendis Pharma Investigational Site, Ivano-Frankivsk
  - Ascendis Pharma Investigational Site, Kharkiv
  - Ascendis Pharma Investigational Site, Kyiv
  - Ascendis Pharma Investigational Site, Vinnytsia
- United Kingdom (3):
  - Ascendis Pharma Investigational Site, Cardiff
  - Ascendis Pharma Investigational Site, Coventry
  - Ascendis Pharma Investigational Site, Leeds

REFERENCES:
- [Derived] Biller BMK, Gilis-Januszewska A, Doknic M, Pico AM, Fleseriu M, Raverot G, Isidori AM, Takahashi Y, Garcia JM, Silverstein JM, Bancos I, Fukuoka H, Huang E, Kang J, Komirenko AS, Domrzalski L, Shu AD, Beckert M, Yuen KCJ. Efficacy and Safety of Once-Weekly Lonapegsomatropin in Adults With Growth Hormone Deficiency: foresiGHt Trial Results. J Clin Endocrinol Metab. 2025 Dec 20:dgaf680. doi: 10.1210/clinem/dgaf680. Online ahead of print. PMID 41420532

RESULTS

PARTICIPANT FLOW:
Groups:
- Lonapegsomatropin: Participants received lonapegsomatropin administered once weekly by subcutaneous injection for a treatment period of up to 38 weeks.
- Placebo: Participants received placebo matched to lonapegsomatropin administered once weekly by subcutaneous injection for a treatment period of up to 38 weeks.
- Somatropin: Participants received somatropin administered once daily by subcutaneous injection for a treatment period of up to 38 weeks.
Period: Overall Study
Arm/Group | Lonapegsomatropin | Placebo | Somatropin
Started | 90 | 87 | 87
Treated | 89 | 84 | 86
Completed | 85 | 81 | 82
Not Completed | 5 | 6 | 5
Not completed — Withdrawal by Subject | 3 | 1 | 2
Not completed — Adverse Event | 1 | 0 | 1
Not completed — Lost to Follow-up | 0 | 1 | 0
Not completed — Physician Decision | 0 | 0 | 1
Not completed — Other | 0 | 1 | 0
Not completed — Randomized but not treated | 1 | 3 | 1

BASELINE CHARACTERISTICS:
Population: Analysis was performed on Intent-to-Treat population that consisted of all randomized participants who received any amount of the trial drug and were analyzed by the treatment arm as randomized.
Groups:
- Total: Total of all reporting groups
Arm/Group | Lonapegsomatropin | Placebo | Somatropin | Total
Number analyzed (Participants) | 89 | 84 | 86 | 259
Age, Continuous [Mean (Standard Deviation); unit: years] | 43.0 (13.40) | 44.1 (14.74) | 41.3 (14.34) | 42.8 (14.15)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 42 | 39 | 38 | 119
  Male | 47 | 45 | 48 | 140
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 3 | 4 | 5 | 12
  Not Hispanic or Latino | 82 | 79 | 78 | 239
  Unknown or Not Reported | 4 | 1 | 3 | 8
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 1 | 0 | 1
  Asian | 11 | 8 | 9 | 28
  Black or African American | 0 | 0 | 1 | 1
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0 | 0
  White | 72 | 71 | 75 | 218
  Other | 6 | 4 | 1 | 11
Dose Group [Count of Participants; unit: Participants]
  Subgroup 1: Oral estrogen intake or <30 years old | 32 | 29 | 30 | 91
  Subgroup 2: >=30 to <=60 years old; no oral estrogen intake | 46 | 43 | 45 | 134
  Subgroup 3: >60 years old; no oral estrogen intake | 11 | 12 | 11 | 34

OUTCOME MEASURES:

1. Primary Outcome: Change From Baseline in Trunk Percent Fat at Week 38
Description: Trunk percent fat was assessed by dual-energy X-ray absorptiometry.
Time Frame: Baseline, Week 38
Population: Analysis was performed on Intent-To-Treat population that consisted of all randomized participants who received any amount of the trial drug and were analyzed by the treatment arm as randomized. Here, "Overall number of participants analyzed" = participants with available data for this outcome measure. Data for this outcome measure was planned to be collected and analyzed for lonapegsomatropin and placebo groups, and not for somatropin group.
Measure: Least Squares Mean (95% Confidence Interval); unit: percent fat
Arm/Group | Lonapegsomatropin | Placebo
Number analyzed (Participants) | 82 | 77
percent fat | -1.68 [-2.44 to -0.91] | 0.37 [-0.30 to 1.03]
Statistical Analysis 1: Comparison: Lonapegsomatropin vs Placebo; Analysis included treatment arm, region, baseline age group, gender, concomitant oral estrogen, Adult Growth Hormone Deficiency (AGHD) onset as factors & baseline trunk percent fat as the covariates. Multiple imputation method was used to impute missing data; Test type: Superiority; p < .0001, ANCOVA; Estimate of Difference = -2.04, 95% CI 2-sided [-2.94 to -1.14], Standard Error of Mean 0.46

2. Secondary Outcome: Change From Baseline in Total Body Lean Mass at Week 38
Description: Total body lean mass was assessed by dual-energy X-ray absorptiometry.
Time Frame: Baseline, Week 38
Population: Analysis was performed on Intent-to-Treat population. Here, "Overall number of participants analyzed" = participants with available data for this outcome measure. Data for this outcome measure was planned to be collected and analyzed for lonapegsomatropin and placebo groups, and not for somatropin group.
Measure: Least Squares Mean (95% Confidence Interval); unit: kilograms
Arm/Group | Lonapegsomatropin | Placebo
Number analyzed (Participants) | 82 | 77
kilograms | 1.60 [1.00 to 2.19] | -0.11 [-0.72 to 0.51]

3. Secondary Outcome: Change From Baseline in Trunk Fat Mass at Week 38
Description: Trunk fat mass was assessed by dual-energy X-ray absorptiometry.
Time Frame: Baseline, Week 38
Population: as for outcome 2
Measure: Least Squares Mean (95% Confidence Interval); unit: kilograms
Arm/Group | Lonapegsomatropin | Placebo
Number analyzed (Participants) | 82 | 77
kilograms | -0.48 [-0.89 to -0.07] | 0.22 [-0.15 to 0.60]

4. Secondary Outcome: Number of Participants With Treatment-Emergent Adverse Events (TEAEs), Serious TEAEs and TEAE Leading to Study Discontinuation
Description: An Adverse Event (AE) is defined as any untoward medical occurrence in a clinical investigation participant administered a pharmaceutical product and which does not necessarily have a causal relationship with the treatment. An AE was considered a TEAE if it occurred on or after the first dose of investigational product and was not present prior to the first dose, or it was present at the first dose but increased in severity during the trial. A serious AE is any untoward medical occurrence at any dose: resulted in death; was life threatening; required prolong inpatient hospitalization; resulted in persistent or significant disability/incapacity; resulted in a congenital anomaly/birth defect or was considered a significant medical event by the investigator.
Time Frame: Up to 38 weeks
Population: Analysis was performed on safety population that included all randomized participants who received any amount of trial drug and was analyzed by the actual treatment received.
Measure: Count of Participants; unit: Participants
Arm/Group | Lonapegsomatropin | Placebo | Somatropin
Number analyzed (Participants) | 89 | 84 | 86
Participants
  TEAEs | 64 | 55 | 63
  Serious TEAEs | 4 | 1 | 6
  TEAE Leading to Study Discontinuation | 1 | 0 | 0

ADVERSE EVENTS:
Time Frame: From signing of the informed consent form (ICF) up to 2 weeks after last dose of the study treatment (i.e., up to Week 40)
Description: Analysis was performed on safety population that included all randomized participants who received any amount of trial drug and was analyzed by the actual treatment received.
Arm/Group | Lonapegsomatropin | Placebo | Somatropin
All-Cause Mortality (participants affected / at risk) | 0/89 | 0/84 | 0/86
Serious Adverse Events (participants affected / at risk) | 4/89 | 1/84 | 6/86
Other Adverse Events (participants affected / at risk) | 29/89 | 47/84 | 28/86
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Lonapegsomatropin (N=89) | Placebo (N=84) | Somatropin (N=86)
Non-cardiac chest pain (General disorders) | 1 (1) | 0 (0) | 0 (0)
Face oedema (General disorders) | 0 (0) | 0 (0) | 1 (1)
Oedema peripheral (General disorders) | 0 (0) | 0 (0) | 1 (1)
Epilepsy (Nervous system disorders) | 1 (1) | 0 (0) | 0 (0)
Seizure (Nervous system disorders) | 0 (0) | 0 (0) | 1 (1)
Coronavirus pneumonia (Infections and infestations) | 1 (1) | 0 (0) | 0 (0)
Hyponatraemia (Metabolism and nutrition disorders) | 1 (1) | 0 (0) | 0 (0)
Acute kidney injury (Renal and urinary disorders) | 0 (0) | 1 (1) | 0 (0)
Anaemia (Blood and lymphatic system disorders) | 0 (0) | 0 (0) | 1 (1)
Transitional cell carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 0 (0) | 1 (1)
Drug eruption (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 1 (1)
Hypertension (Vascular disorders) | 0 (0) | 0 (0) | 1 (1)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Lonapegsomatropin (N=89) | Placebo (N=84) | Somatropin (N=86)
COVID-19 (Infections and infestations) | 7 (7) | 11 (11) | 6 (7)
Arthralgia (Musculoskeletal and connective tissue disorders) | 8 (8) | 8 (8) | 7 (9)
Nasopharyngitis (Infections and infestations) | 5 (6) | 11 (16) | 6 (7)
Headache (Nervous system disorders) | 7 (13) | 9 (11) | 5 (5)
Upper respiratory tract infection (Infections and infestations) | 2 (2) | 8 (10) | 4 (5)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (2):
  • Study Protocol (2022-06-02): https://cdn.clinicaltrials.gov/large-docs/73/NCT04615273/Prot_000.pdf
  • Statistical Analysis Plan (2023-11-01): https://cdn.clinicaltrials.gov/large-docs/73/NCT04615273/SAP_001.pdf